CLINICAL TRIAL: NCT01667965
Title: Use of a Video Decision Tool to Improve Informed Decision-Making in Hospitalized Patients Considering Palliative Radiation Therapy
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 12-172
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Metastatic Cancer or Locally Advanced; Patients Receiving Palliative Radiation
Keywords: palliative radiation; 12-172
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- pts receiving palliative radiation therapy: The design of the study will be a prospective non-randomized cohort study with structured questionnaires administered to all enrolled patients at two or three time-points.
  Interventions: Behavioral: questionnaires

INTERVENTIONS:
Behavioral: questionnaires — Questionnaires will be given before the patient watches a video educational tool to aid informed consent about palliative radiation therapy; and (2) after the patient watches the video educational tool. (3) If the patient receives PRT, a final questionnaire that assesses the patient's impression of the video will also be administered at the conclusion of radiation therapy.

SUMMARY:
The purpose of this study is to assess the effectiveness and acceptability of a recently created informative video geared for patients who have been evaluated by a radiation oncologist for palliative radiation therapy during a hospitalization at Memorial Sloan-Kettering Cancer Center. Palliative radiation therapy is radiation therapy that is given to patients with the purpose of easing symptoms from cancer. It is not given with the intent to cure the cancer. The video presents basic information about palliative radiation and palliative care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Eligible for palliative radiation to the brain, spine, chest, abdomen, pelvis, skin, or bone as per the judgment of the radiation oncologist or nurse practitioner
* Patient is English-speaking and able to give informed consent and fill out study questionnaires
* Hospitalized at MSKCC
* Pathologically confirmed malignancy
* Cancer is metastatic or locally advanced, and is not curable
* Patients who may undergo radiation at a satellite facility are still eligible for protocol enrollment

Exclusion Criteria:

* Those who have seen the video beforehand

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients will be approached regarding study enrollment at the time that they are evaluated by the inpatient radiation oncology team for palliative radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2012-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
create an effective video decision aid | 1 year
  Effectiveness of the video tool will be assessed by the following measures before and after watching the video. The pre- and post-assessment design comparing uncertainty, knowledge and preference scores of a video explaining palliative radiation and palliative care.

CONTACTS AND LOCATIONS:
Overall Officials: Beryl McCormack, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/